CLINICAL TRIAL: NCT07108556
Title: Brief Mindfulness Workshop With or Without Virtual Reality: A Randomized Crossover Design
Brief Title: Brief Mindfulness Workshop With or Without Virtual Reality: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: New Life Psychiatric Rehabilitation Association (Other)
Responsible Party: Principal Investigator, Amanda Kingsze CHEUNG, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EA250376
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mental Wellbeing

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Add-on (with VR-incorporated first) (Experimental): Mindfulness exercise with virtual reality incorporated as the first experiential session
  Interventions: Behavioral: Mindfulness VR-Typical
- Mindfulness Typical (audio-only first) (Active Comparator): Mindfulness exercise with only audio guidance as the first experiential session
  Interventions: Behavioral: Mindfulness Typical-VR

INTERVENTIONS:
Behavioral: Mindfulness VR-Typical — Participants first experience mindfulness exercise with virtual reality incorporated, then another mindfulness exercise with only audio-guidance as typically delivered without the technology
  Arms: Mindfulness Add-on (with VR-incorporated first)
Behavioral: Mindfulness Typical-VR — Participants first experience mindfulness exercise with only audio-guidance, then another mindfulness exercise with virtual reality incorporated
  Arms: Mindfulness Typical (audio-only first)

SUMMARY:
The current study uses a randomized cross-over design, in which participants are exposed to brief mindfulness-based experiential sessions with and without incorporating virtual reality (i.e., the experimental and control conditions, respectively). Order of exposure to these two conditions are counter-balanced and participants are randomized into the two arms of exposure in a different order. Furthermore, this study includes the use of both subjective self-report and objective physiological measures of mental wellbeing. It is hypothesized that VR-incorporated mindfulness-based experiential session brings a greater improvement in state mindfulness, state affect, and stress response. Results shed light on the added value of incorporating VR into brief MBIs, particularly in reference to the typical practice of promoting mindfulness in the local community.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* reads Chinese
* understands Cantonese

Exclusion Criteria:

* history of sever motion sickness or known intolerance to VR environments
* impairments that may interfere with the use of VR equipment
* concurrent or past structured mindfulness training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in positive affect as measured by International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) after a brief practice of mindfulness. | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  Using a 5-point Likert scale from 1 = Never to 5 = Always, individuals rate on their experience of five positive affect in the present moment. Scores are summed across 5 items, with higher scores indicating higher levels of positive affect.
Change in negative affect as measured by International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) after a brief practice of mindfulness. | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  Using a 5-point Likert scale from 1 = Never to 5 = Always, individuals rate on their experience of five negative affect in the present moment. Scores are summed across 5 items, with higher scores indicating higher levels of negative affect.
Change in state mindfulness as measured by the State Mindfulness Scale (SMS) after a brief practice of mindfulness. | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  Individuals rate their state mindfulness on a 5-point Likert scale across 21 items, from 1 = Not at All to 5 = Very Much. Scores are summed to represent overall mindfulness and two subfactors differentiated by objects of mindfulness - (1) mind and (2) body. Higher scores indicate higher levels of mindfulness at the moment.
Change in heart rate variability as measured with the Shimmer3 GSR+ (Galvanic Skin Response) unit after a brief practice of mindfulness. | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  The Shimmer3 GSR+ unit is strapped to a participant's wrist and fingers of the non-dominant hand. An optical pulse sensor is attached to the second finger to collect photoplethysmogram (PPG) signals over a 5-minute period, which are then transformed into HRV measures with artifacts corrected through automated detection using the Kubios HRV Scientific software. Higher values indicate greater heart rate variability.
Change in skin conductance level as measured with the Shimmer3 GSR+ (Galvanic Skin Response) unit after a brief practice of mindfulness. | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  The Shimmer3 GSR+ unit is strapped to a participant's wrist and fingers of the non-dominant hand. Two additional electrodes are attached to the third and fourth fingers of the participants' non-dominant hand to collect both phasic and tonic skin conductance data. Higher values indicate greater skin conductance.

SECONDARY OUTCOMES:
Satisfaction with the intervention as measured by a single Likert item with open text entry designed specifically for this study | At the end of the full program (i.e., one-time assessment; at minute 20).
  Participants complete a service evaluation form that includes rating on a 5-point Likert scale, from 1 - Strongly Disagree to 5 - Strongly Agree, designed specifically to assess their level of satisfaction with the intervention received in the current study. They are also asked in an open-ended way to provide narratives of their experience throughout the encounter.

OTHER OUTCOMES:
Level of engagement or presence during a mindfulness exercise as measured by 3-5 Likert items designed specifically for this study | At the start of the first session (at minute 0), at the end of the first session (which is also the start of the second session; at minute 10), and at the end of the second session (at minute 20).
  Using a 5-point Likert scale, from 1 - Strongly Disagree to 5 - Strongly Agree, all participants rate on 3 items that assess their engagement, sense of being, and distractedness during a session. Two more items are to be completed if VR technology is involved in the experiential session.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Cheung, Principal Investigator — The University of Hong Kong
Locations (1):
- New Life Psychiatric Rehabilitation Association, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Not covered in informed consent